CLINICAL TRIAL: NCT02326155
Title: An Observational, Prospective Cohort Study to Evaluate the Safety and Efficacy of Remsima™ in Patients With Crohn's Disease (CD) or Ulcerative Colitis (UC)
Brief Title: To Evaluate the Safety and Efficacy of Remsima™ in Patients With Crohn's Disease (CD) or Ulcerative Colitis (UC)
Status: Terminated | Type: Observational
Why Stopped: Terminated
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-P13 4.3
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Results first posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-12

CONDITIONS: Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Remsima™: Patients were not treated with infliximab before enrollment. Patients were administered CT-P13 5mg/kg by intravenous infusion at weeks 0, 2, and 6, and every 8 weeks thereafter.
- Switched to Remsima: Patients were treated with infliximab prior to enrollment of the study. Patients were administered CT-P13 5mg/kg by intravenous infusion at weeks 0, 2, and 6, and every 8 weeks thereafter.

SUMMARY:
An observational, prospective cohort study to evaluate the safety and efficacy of Remsima™ in patients with Crohn's disease (CD) or Ulcerative Colitis (UC)

DETAILED DESCRIPTION:
This is a longitudinal, observational, prospective cohort study to assess the safety and efficacy of Remsima™ in patients with IBD, who have active Crohn's disease (CD), fistulizing Crohn's disease (CD), or Ulcerative Colitis (UC). Patients will be included in this registry who are receiving treatment with 5 mg/kg of Remsima™ by IV infusion at weeks 0, 2, 6, and every 8 weeks thereafter in accordance with the product label. If a patient has been treated with infliximab prior to enrollment, his or her dosing schedule will be continued appropriately. Patients will undergo safety and efficacy assessments in accordance with routine medical practice. The decision to treat with RemsimaTM will be independent of the decision to enroll the patient in this registry.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with moderate to severe active CD
* Children and adolescent patients, aged 6 to 17 years old with severe active CD
* Adult patients with fistulizing active CD
* Adult patients with moderate to severe active UC
* Female patients of childbearing potential who agree to use of adequate contraception to prevent pregnancy and continuation of contraceptive use for at least 6 months after their final dose of Remsima™.
* Patients (or legal guardian, if applicable) who are willing to give informed consent for long term follow-up including access to all medical records.

Exclusion Criteria:

* Patients with a history of hypersensitivity to infliximab
* Patients with a current or past history of chronic infection
* Patients with current diagnosis of Tuberculosis (TB) or severe or chronic infections (e.g. sepsis, abscesses, opportunistic infections, invasive fungal infections), or previously diagnosed with TB or severe or chronic infection, without sufficient documentation of complete resolution following treatment.
* Recent exposure to persons with active TB, or a positive test result for latent TB (determined by a positive interferon-γ release assay [IGRA] test, with a negative chest X-ray) at Screening
* Patients with moderate or severe heart failure (NYHA class III/IV).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of at least 500 male and female patients with active CD, fistulizing active CD, and UC
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Svoboda, Principal Investigator — Ostrava, Morvskoslezsky kraj, Czech Republic, 708 52

REFERENCES:
- [Derived] Cheon JH, Nah S, Kang HW, Lim YJ, Lee SH, Lee SJ, Kim SH, Jung NH, Park JE, Lee YJ, Jeon DB, Lee YM, Kim JM, Park SH. Infliximab Biosimilar CT-P13 Observational Studies for Rheumatoid Arthritis, Inflammatory Bowel Diseases, and Ankylosing Spondylitis: Pooled Analysis of Long-Term Safety and Effectiveness. Adv Ther. 2021 Aug;38(8):4366-4387. doi: 10.1007/s12325-021-01834-3. Epub 2021 Jul 12. PMID 34250583

RESULTS

PARTICIPANT FLOW:
Groups:
- Remsima (CT-P13): Patients were not treated with infliximab before enrollment. Patients were administered CT-P13 5mg/kg by intravenous infusion at weeks 0, 2, and 6, and every 8 weeks thereafter.
- Switched to Remsima (CT-P13): Patients were treated with infliximab prior to enrollment of the study. Patients were administered CT-P13 5mg/kg by intravenous infusion at weeks 0, 2, and 6, and every 8 weeks thereafter.
Period: Overall Study
Arm/Group | Remsima (CT-P13) | Switched to Remsima (CT-P13)
Started | 407 | 63
Completed | 13 | 1
Not Completed | 394 | 62
Not completed — Adverse Event | 21 | 5
Not completed — Death | 3 | 0
Not completed — Lack of Efficacy | 49 | 5
Not completed — Lost to Follow-up | 14 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 34 | 11
Not completed — Disease progression | 37 | 4
Not completed — Study close | 188 | 21
Not completed — except for study close | 46 | 13

BASELINE CHARACTERISTICS:
Population: Safety analysis set, consist of all patients who received at least one dose of the study treatment during any dosing period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Remsima (CT-P13) | Switched to Remsima (CT-P13) | Total
Number analyzed (Participants) | 407 | 63 | 470
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52 | 18 | 70
  Between 18 and 65 years | 334 | 44 | 378
  >=65 years | 21 | 1 | 22
Age, Continuous [Median (Full Range); unit: years] | 33 [8 to 81] | 27 [7 to 69] | 32 [7 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 21 | 190
  Male | 238 | 42 | 280
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 186 | 30 | 216
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 220 | 33 | 253
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Patients Who Experienced Adverse Events of Special Interest (AESI)
Description: Including Hepatitis B virus (HBV) reactivation, congestive heart failure, opportunistic infections (excluding tuberculosis), serious infections including sepsis (excluding opportunistic infections and tuberculosis), tuberculosis (TB), serum sickness (delayed hypersensitivity reactions), haematologic reactions, systemic lupus erythematosus/lupus-like syndrome, demyelinating disorders, lymphoma (not hepatosplenic T cell lymphoma), hepatobiliary events, hepatosplenic T cell lymphoma, intestinal or perianal abscess (in Crohn's disease), serious infusion reactions during a re-induction regimen following disease flare, sarcoidosis/sarcoid-like reactions, paediatric malignancy, leukaemia, malignancy (excluding lymphoma), colon carcinoma/dysplasia (in Ulcerative Colitis), skin cancer, pregnancy exposure, bowel stenosis/stricture/obstruction (in Crohn's disease) and infusion related reaction (IRR)/ hypersensitivity/anaphylactic reaction.
Time Frame: Up to 5 years for each patient
Population: Safety analysis set, all patients who received at least one dose of study treatment. Intestinal or perianal abscess and bowel stenosis/stricture/obstruction events are only applicable for patients with moderate to severe active CD, fistulising active CD and paediatric severe active CD. Colon carcinoma/dysplasia is only applicable for patients with moderate to severe active UC and paediatric severe active UC. Paediatric malignancy is only applicable for paediatric patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Remsima (CT-P13) | Switched to Remsima (CT-P13)
Number analyzed (Participants) | 407 | 63
Participants
  Treatment-emergent Adverse Events (TEAEs) of Hepatitis B virus reactivation | 0 | 0
  Treatment-emergent Adverse Events of congestive heart failure | 0 | 0
  Treatment-emergent Adverse Events of opportunistic infections (excluding tuberculosis) | 0 | 0
  TEAEs of serious infections including sepsis (excl. opportunistic infections and TB | 15 | 2
  Treatment-emergent Adverse Events of tuberculosis (TB) | 4 | 0
  Treatment-emergent Adverse Events of serum sickness (delayed hypersensitivity reactions) | 0 | 0
  Treatment-emergent Adverse Events of haematologic reactions | 36 | 8
  Treatment-emergent Adverse Events of systemic lupus erythematosus/lupus-like syndrome | 0 | 0
  Treatment-emergent Adverse Events of demyelinating disorders | 0 | 0
  Treatment-emergent Adverse Events of lymphoma (not hepatosplenic T cell lymphoma) | 1 | 0
  Treatment-emergent Adverse Events of hepatobiliary events | 14 | 5
  Treatment-emergent Adverse Events of hepatosplenic T cell lymphoma | 0 | 0
  Treatment-emergent Adverse Events of intestinal or perianal abscess (in Crohn's disease): number analyzed (Participants) | 250 | 53
  Treatment-emergent Adverse Events of intestinal or perianal abscess (in Crohn's disease) | 7 | 1
  TEAEs of serious infusion reactions during a re-induction regimen following disease flare | 0 | 0
  Treatment-emergent Adverse Events of sarcoidosis/sarcoid-like reactions | 0 | 1
  Treatment-emergent Adverse Events of paediatric malignancy: number analyzed (Participants) | 47 | 15
  Treatment-emergent Adverse Events of paediatric malignancy | 0 | 0
  Treatment-emergent Adverse Events of leukaemia | 0 | 0
  Treatment-emergent Adverse Events of malignancy (excluding lymphoma) | 3 | 2
  Treatment-emergent Adverse Events of colon carcinoma/dysplasia (in Ulcerative Colitis): number analyzed (Participants) | 157 | 10
  Treatment-emergent Adverse Events of colon carcinoma/dysplasia (in Ulcerative Colitis) | 0 | 0
  Treatment-emergent Adverse Events of skin cancer | 0 | 0
  Treatment-emergent Adverse Events of pregnancy exposure | 3 | 1
  Treatment-emergent Adverse Events of bowel stenosis/stricture/obstruction (in Crohn's disease): number analyzed (Participants) | 250 | 53
  Treatment-emergent Adverse Events of bowel stenosis/stricture/obstruction (in Crohn's disease) | 8 | 2
  TEAEs of infusion related reaction (IRR)/ hypersensitivity/anaphylactic reaction | 39 | 4

2. Secondary Outcome: Number and Percentage of Patients Achieving Clinical Response, Decrease of ≥70 Points From Baseline Scores in Crohn's Disease Activity Index-70 (CDAI-70) and Decrease of ≥100 Points From Baseline Scores in CDAI-100
Description: A patient is considered as achieving clinical response according to CDAI-70 (or CDAI-100) if the patient has a reduction on CDAI score of 70 (or 100) points or more from the baseline value.
Time Frame: Every 6 months (months 6 -60)
Population: Efficacy analysis set, consist of all moderate-severe active Crohn's Disease patients who received at least one dose of the study treatment during any dosing period and had at least one efficacy result corresponding to indication used for analysis after treatment. The denominators of proportions are the number of patients with non-missing efficacy result at each time point and baseline. Some rows have 0 participants analyzed because there were no patients applicable for analysis on this visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Remsima (CT-P13) | Switched to Remsima (CT-P13)
Number analyzed (Participants) | 124 | 23
Participants
  Clinical response according to CDAI-70 at 6 months: number analyzed (Participants) | 68 | 14
  Clinical response according to CDAI-70 at 6 months | 36 | 2
  Clinical response according to CDAI-70 at 12 months: number analyzed (Participants) | 69 | 15
  Clinical response according to CDAI-70 at 12 months | 42 | 4
  Clinical response according to CDAI-70 at 18 months: number analyzed (Participants) | 68 | 11
  Clinical response according to CDAI-70 at 18 months | 39 | 3
  Clinical response according to CDAI-70 at 24 months: number analyzed (Participants) | 47 | 13
  Clinical response according to CDAI-70 at 24 months | 27 | 4
  Clinical response according to CDAI-70 at 30 months: number analyzed (Participants) | 38 | 9
  Clinical response according to CDAI-70 at 30 months | 24 | 0
  Clinical response according to CDAI-70 at 36 months: number analyzed (Participants) | 28 | 4
  Clinical response according to CDAI-70 at 36 months | 22 | 0
  Clinical response according to CDAI-70 at 42 months: number analyzed (Participants) | 22 | 3
  Clinical response according to CDAI-70 at 42 months | 13 | 0
  Clinical response according to CDAI-70 at 54 months: number analyzed (Participants) | 16 | 4
  Clinical response according to CDAI-70 at 54 months | 12 | 0
  Clinical response according to CDAI-70 at 48 months: number analyzed (Participants) | 9 | 1
  Clinical response according to CDAI-70 at 48 months | 8 | 0
  Clinical response according to CDAI-70 at 60 months: number analyzed (Participants) | 2 | 0
  Clinical response according to CDAI-70 at 60 months | 2 |
  Clinical response according to CDAI-100 at 6 months: number analyzed (Participants) | 68 | 14
  Clinical response according to CDAI-100 at 6 months | 33 | 2
  Clinical response according to CDAI-100 at 12 months: number analyzed (Participants) | 69 | 15
  Clinical response according to CDAI-100 at 12 months | 36 | 3
  Clinical response according to CDAI-100 at 18 months: number analyzed (Participants) | 68 | 11
  Clinical response according to CDAI-100 at 18 months | 34 | 3
  Clinical response according to CDAI-100 at 24 months: number analyzed (Participants) | 47 | 13
  Clinical response according to CDAI-100 at 24 months | 24 | 2
  Clinical response according to CDAI-100 at 30 months: number analyzed (Participants) | 38 | 9
  Clinical response according to CDAI-100 at 30 months | 24 | 0
  Clinical response according to CDAI-100 at 36 months: number analyzed (Participants) | 28 | 4
  Clinical response according to CDAI-100 at 36 months | 18 | 0
  Clinical response according to CDAI-100 at 42 months: number analyzed (Participants) | 22 | 3
  Clinical response according to CDAI-100 at 42 months | 12 | 0
  Clinical response according to CDAI-100 at 48 months: number analyzed (Participants) | 16 | 4
  Clinical response according to CDAI-100 at 48 months | 12 | 0
  Clinical response according to CDAI-100 at 54 months: number analyzed (Participants) | 9 | 1
  Clinical response according to CDAI-100 at 54 months | 8 | 0
  Clinical response according to CDAI-100 at 60 months: number analyzed (Participants) | 2 | 0
  Clinical response according to CDAI-100 at 60 months | 2 |

3. Secondary Outcome: Number and Percentage of Patients Achieving Clinical Response, Decrease From Baseline in the Paediatric Crohn's Disease Activity Index (PCDAI) ≥15 Points; Total Score ≤30
Description: A patient is considered as achieving clinical response according to PCDAI if the patient has a PCDAI score less than or equal to 30 points and a reduction on PCDAI score of 15 points or more from the baseline value.
Time Frame: Every 6 months (months 6 -42)
Population: Efficacy analysis set, consist of all Pediatric severe active Crohn's Disease patients who received at least one dose of the study treatment during any dosing period and had at least one efficacy result corresponding to indication used for analysis after treatment. The denominators of proportions are the number of patients with non-missing efficacy result at each timepoint and baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Remsima (CT-P13) | Switched to Remsima (CT-P13)
Number analyzed (Participants) | 41 | 15
Participants
  Clinical response at 6 months: number analyzed (Participants) | 32 | 11
  Clinical response at 6 months | 15 | 2
  Clinical response at 12 months: number analyzed (Participants) | 35 | 13
  Clinical response at 12 months | 18 | 2
  Clinical response at 18 months: number analyzed (Participants) | 31 | 9
  Clinical response at 18 months | 17 | 0
  Clinical response at 24 months: number analyzed (Participants) | 22 | 9
  Clinical response at 24 months | 10 | 0
  Clinical response at 30 months: number analyzed (Participants) | 6 | 3
  Clinical response at 30 months | 0 | 0
  Clinical response at 36 months: number analyzed (Participants) | 6 | 7
  Clinical response at 36 months | 2 | 1
  Clinical response at 42 months: number analyzed (Participants) | 6 | 8
  Clinical response at 42 months | 1 | 1

4. Secondary Outcome: Number and Percentage of Patients Achieving Clinical Response, a ≥50% Reduction From Baseline in the Number of Draining Fistulas Over a Period of ≥4 Weeks Compared to Baseline
Description: A patient is considered as achieving clinical response according to the number of draining fistulas if the patient has a reduction on the number of draining fistulas from the baseline value (over a period of ≥ 4 weeks) ≥ 50%.
Time Frame: Every 6 months (months 6 -48)
Population: Efficacy analysis set, consist of all Fistulizing Active Crohn's Disease patients who received at least one dose of the study treatment during any dosing period and had at least one efficacy result corresponding to indication used for analysis after treatment. The denominators of proportions are the number of patients with non-missing efficacy result at each timepoint and baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Remsima (CT-P13) | Switched to Remsima (CT-P13)
Number analyzed (Participants) | 19 | 6
Participants
  Clinical response at 6 months: number analyzed (Participants) | 14 | 6
  Clinical response at 6 months | 2 | 1
  Clinical response at 12 months: number analyzed (Participants) | 12 | 5
  Clinical response at 12 months | 3 | 1
  Clinical response at 18 months: number analyzed (Participants) | 8 | 3
  Clinical response at 18 months | 4 | 0
  Clinical response at 24 months: number analyzed (Participants) | 4 | 2
  Clinical response at 24 months | 2 | 0
  Clinical response at 30 months: number analyzed (Participants) | 3 | 1
  Clinical response at 30 months | 2 | 0
  Clinical response at 36 months: number analyzed (Participants) | 2 | 2
  Clinical response at 36 months | 1 | 0
  Clinical response at 42 months: number analyzed (Participants) | 1 | 1
  Clinical response at 42 months | 0 | 1
  Clinical response at 48 months: number analyzed (Participants) | 1 | 1
  Clinical response at 48 months | 0 | 1

5. Secondary Outcome: Decrease in Mayo Scores From Baseline at Least 3 Points and 30% for Total or Decrease in Scores From Baseline at Least 2 Points for Partial, With Accompanying Decrease in Subscore for Rectal Bleeding of at Least 1 Point, or Absolute Subscore 0 or 1.
Description: A patient is considered as achieving clinical response according to total Mayo score if the patient has a reduction from baseline in total mayo score at least 3 points and at least 30%, with an accompanying reduction in the subscore for rectal bleeding of at least 1 point, or an absolute subscore for rectal bleeding of 0 or 1. A patient is considered as achieving clinical response according to partial Mayo score if the patient has a reduction from baseline in partial mayo score at least 2 points, with an accompanying reduction in the subscore for rectal bleeding of at least 1 point, or an absolute subscore for rectal bleeding of 0 or 1.
Time Frame: Every 6 months (months 6 - 60)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Remsima (CT-P13) | Switched to Remsima (CT-P13)
Number analyzed (Participants) | 103 | 6
Participants
  Clinical response according to total mayo score at 6 months: number analyzed (Participants) | 34 | 0
  Clinical response according to total mayo score at 6 months | 18 |
  Clinical response according to total mayo score at 12 months: number analyzed (Participants) | 31 | 0
  Clinical response according to total mayo score at 12 months | 19 |
  Clinical response according to total mayo score at 18 months: number analyzed (Participants) | 22 | 0
  Clinical response according to total mayo score at 18 months | 13 |
  Clinical response according to total mayo score at 24 months: number analyzed (Participants) | 18 | 0
  Clinical response according to total mayo score at 24 months | 12 |
  Clinical response according to total mayo score at 30 months: number analyzed (Participants) | 18 | 0
  Clinical response according to total mayo score at 30 months | 15 |
  Clinical response according to total mayo score at 36 months: number analyzed (Participants) | 8 | 1
  Clinical response according to total mayo score at 36 months | 5 | 0
  Clinical response according to total mayo score at 42 months: number analyzed (Participants) | 8 | 0
  Clinical response according to total mayo score at 42 months | 7 |
  Clinical response according to total mayo score at 48 months: number analyzed (Participants) | 7 | 0
  Clinical response according to total mayo score at 48 months | 6 |
  Clinical response according to total mayo score at 54 months: number analyzed (Participants) | 5 | 0
  Clinical response according to total mayo score at 54 months | 4 |
  Clinical response according to total mayo score at 60 months: number analyzed (Participants) | 1 | 0
  Clinical response according to total mayo score at 60 months | 1 |
  Clinical response according to partial mayo score at 6 months: number analyzed (Participants) | 54 | 1
  Clinical response according to partial mayo score at 6 months | 35 | 1
  Clinical response according to partial mayo score at 12 months: number analyzed (Participants) | 48 | 2
  Clinical response according to partial mayo score at 12 months | 30 | 1
  Clinical response according to partial mayo score at 18 months: number analyzed (Participants) | 41 | 2
  Clinical response according to partial mayo score at 18 months | 28 | 1
  Clinical response according to partial mayo score at 24 months: number analyzed (Participants) | 33 | 3
  Clinical response according to partial mayo score at 24 months | 22 | 1
  Clinical response according to partial mayo score at 30 months: number analyzed (Participants) | 28 | 1
  Clinical response according to partial mayo score at 30 months | 23 | 1
  Clinical response according to partial mayo score at 36 months: number analyzed (Participants) | 23 | 2
  Clinical response according to partial mayo score at 36 months | 19 | 1
  Clinical response according to partial mayo score at 42 months: number analyzed (Participants) | 18 | 2
  Clinical response according to partial mayo score at 42 months | 15 | 1
  Clinical response according to partial mayo score at 48 months: number analyzed (Participants) | 15 | 2
  Clinical response according to partial mayo score at 48 months | 14 | 1
  Clinical response according to partial mayo score at 54 months: number analyzed (Participants) | 12 | 0
  Clinical response according to partial mayo score at 54 months | 10 |
  Clinical response according to partial mayo score at 60 months: number analyzed (Participants) | 2 | 0
  Clinical response according to partial mayo score at 60 months | 2 |

6. Secondary Outcome: Number and Percentage of Patients Achieving Clinical Response, Decrease From Baseline in the Paediatric Ulcerative Colitis Activity Index (PUCAI) ≥20 Score
Description: A patient is considered as achieving clinical response according to PUCAI if the patient has a reduction on PUCAI score of 20 points or more from the baseline value.
Time Frame: Every 6 months (months 6 - 18)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Remsima (CT-P13) | Switched to Remsima (CT-P13)
Number analyzed (Participants) | 2 | 0
Participants
  Clinical response at 6 months | 1 |
  Clinical response at 12 months | 1 |
  Clinical response at 18 months: number analyzed (Participants) | 1 | 0
  Clinical response at 18 months | 1 |

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date the patient signed the informed consent form and until the end of study visit up to 5 years, an average of 26.345 months. .
Arm/Group | Remsima (CT-P13) | Switched to Remsima (CT-P13)
All-Cause Mortality (participants affected / at risk) | 5/407 | 0/63
Serious Adverse Events (participants affected / at risk) | 53/407 | 10/63
Other Adverse Events (participants affected / at risk) | 221/407 | 34/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remsima (CT-P13) (N=407) | Switched to Remsima (CT-P13) (N=63)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileal stenosis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0
Large intestinal perforation (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Generalised Oedema (General disorders) | 1 | 0
Localised Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Chronic Hepatitis B (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 0
Rotavirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
High risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal infarct (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remsima (CT-P13) (N=407) | Switched to Remsima (CT-P13) (N=63)
Anaemia (Blood and lymphatic system disorders) | 17 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 2
Vision blurred (Eye disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 56 | 9
Abdominal pain upper (Gastrointestinal disorders) | 13 | 1
Anal fissure (Gastrointestinal disorders) | 3 | 2
Anal fistula (Gastrointestinal disorders) | 6 | 3
Anal inflammation (Gastrointestinal disorders) | 0 | 3
Anal skin tags (Gastrointestinal disorders) | 0 | 3
Aphthous ulcer (Gastrointestinal disorders) | 1 | 6
Cheilosis (Gastrointestinal disorders) | 1 | 2
Colitis ulcerative (Gastrointestinal disorders) | 16 | 0
Crohn's disease (Gastrointestinal disorders) | 48 | 11
Diarrhoea (Gastrointestinal disorders) | 37 | 11
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 11 | 3
Gastritis (Gastrointestinal disorders) | 10 | 2
Gastrooesophagel reflux disease (Gastrointestinal disorders) | 5 | 2
Haematochezia (Gastrointestinal disorders) | 21 | 6
Ileal stenosis (Gastrointestinal disorders) | 1 | 2
Mucous stools (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 17 | 4
Vomiting (Gastrointestinal disorders) | 18 | 3
Asthenia (General disorders) | 13 | 4
Pyrexia (General disorders) | 18 | 4
Hypertransaminaesaemia (Hepatobiliary disorders) | 1 | 2
Bacteriuria (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 41 | 7
Oral herpes (Infections and infestations) | 12 | 2
Pharyngitis (Infections and infestations) | 17 | 6
Rhinitis (Infections and infestations) | 13 | 5
Upper respiratory tract infection (Infections and infestations) | 24 | 7
Urinary tract infection (Infections and infestations) | 6 | 2
Varicella zoster virus infection (Infections and infestations) | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 32 | 4
Bone density decreased (Investigations) | 5 | 5
Faecal calprotectin increased (Investigations) | 3 | 6
Hepatic enzyme increased (Investigations) | 2 | 2
Red blood cell sedimentation rate increased (Investigations) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Dizziness (Nervous system disorders) | 15 | 2
Headache (Nervous system disorders) | 24 | 4
Mood swings (Psychiatric disorders) | 7 | 2
Dysuria (Renal and urinary disorders) | 1 | 2
Leukocyturia (Renal and urinary disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Acne (Skin and subcutaneous tissue disorders) | 12 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-06-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT02326155/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT02326155/SAP_001.pdf